1 2

Blood Loss Reduction After Total Knee Arthroplasty. Comparison Topical Tranexamic Acid vs Platelet Rich Plasma

NCT02650856

6 Document Date: October 21, 2019 7 Date of Study Closure: April 26 2017

## Statistical analysis Plan

The sample size was calculated using the following characteristics: 90% power and a critical p value of 0.05 for a decrease in the transfusion rate of 100% based on a previous report and on the assumption that may abate transfusion requirements.[21] This resulted in a total of 40 patients. Central tendency and dispersion measures were calculated for the numerical variables, and frequencies and percentages were calculated for the categorical variables. The Kolmogorov-Smirnov test was performed to test the normal distribution of all numerical variables. In the case of parametric numerical variables, Student's t-tests, one-way ANOVA, and multiple comparisons ANOVA were performed for related and independent samples. For non-parametric numerical variables, Mann-Whitney U, Wilcoxon, and Kruskal Wallis tests were performed. The Bonferroni sequential correction test was performed in the post hoc analyses. Statistical significance was set at a value of p < 0.05. The SPSS version 20.0 (IBM, Armonk, NY) statistical package for Windows 7 was used for the statistical analysis.

## **Brief Summary**

- The investigators will include patients who will be schedule for total knee
- 26 arthroplasty with a diagnosis of osteoarthritis. The patients will be divided in two

groups. In both groups a verbal and clear detailed information will be given on the intraoperative approach. The first group will receive topical tranexamic acid and the second group topical platelet rich plasma; both in the surgical site. Both groups will be assessed before and after the intervention with laboratory results (hemoglobin, hematocrit levels) and drainage drain.

## **Detailed Description:**

27

28

29

30

31

32

33

34

35

36

37

38

39

40

41

42

43

44

45

46

47

48

49

50

Total knee replacement (TKR) surgery is one the most common orthopaedic procedure in the world. Morbility in perioperative TKR is associated to: blood loss, pain, infection, wound complications, stiffness and thrombotic events. Blood loss and transfusion have been associated to increased hospital stay, costs, morbility and mortality of the patient. Indications for blood transfusions are now limited and it is well known that is not a free risk procedure. Complications such as; ABO incompatibility, viral transmission, hemolysis, immunosuppression and wound infection have been reported. Literature reports have reported blood loss in TKR ranging from 300ml to 1 liter, and transfusion rate varying from 10-38%. In diminishing hospital cost Moskal J. et al reported 53.90% of savings and a 100% reduction in working hours of the hospital staff using topical tranexamic acid in TKR. Tranexamic acid is an antifibrinolytic agent that acts inhibiting the plasminogen, stabilizing the blood clot; it is used to stop surgical or traumatic bleeding like in the CRASH-2 trial, demonstrating its efficiency in the polytraumatized patients. Tranexamic acid has been used in the last years for blood loss with good results. Due to its systemic effects and past medical history of myocardial infarction, stents and previous thromboembolic events its intravenous use is limited. In this study the investigators

- will use topical tranexamic acid and its use has been proven in clinical trials as
- 52 secure strategy por blood loss reduction in TKR, without excluding patients with
- 53 previous thromboembolic events.
- Platelet rich plasma (PRP) is an orthobiologic that has played an important role
- over the past decade in different areas like; spinal fusion, ACL reconstruction,
- osteoarthrosis and tendinopathies. The use of platelet rich plasma (PRP) in
- orthopaedics is overrated and true indications for its use and cost benefit are still
- unclear. Retrospective studies like Pace T et al in 268 patients did not
- 59 demonstrated differences in hospital stay, Postoperative hemoglobin levels, range
- of motion with the use PRP in TKR. Morishita M. Et al in a clinical trial of 40
- patients, using intralesional PRP didn't show any benefits for blood loss reduction
- in TKR, but good clinical results were observed in clinical scores like KOOS and
- VAS compared to the control group. Other studies have demonstrated the efficacy
- of topical PRP in blood loss reduction in TKR.
- Due to its high platelet concentration and growth factors contained in the alfa
- granules; it is used as an hemostatic, analgesic and antiseptic agent in TKR.
- 67 There is a variety of blood loss prevention strategies for TKR and this strategies
- can be divided in preoperative, intraoperative or postoperative. The aim of this
- study is to compare the use of topical tranexamic acid versus topical platelet rich
- 70 plasma.
- An Insall knee approach, parapatellar medial will be used in all the patients. After
- the final cuts of the femoral, tibial and patellar and before placing the final
- cemented components the experimental intervention of the study will begin.
- Group 1. A dosis of 2 gr of tranexamic acid (1000mg/10mL X-GEN

- 75 pharmaceuticals inc.) is diluted in 80mL of physiologic solution and will be divided
- in two applications:
- 77 First application: 40mL of the solution previously prepared is applied over the
- surgical site and it will be left for five minutes then drained out completely by
- 79 suction.
- 80 Second application: The rest of 40mL of solution previously prepared is applied
- after placing the final TKR cemented components (femoral, tibial and patellar), over
- the surgical site and leaving it there without draining it by suction.
- 83 Group 2. In the preoperative room with previous premedication, a total of 55cc of
- total venous blood is obtained from the forearm (cubital o basilic veins). The blood
- is carried on 12 steriles tubes using sodium citrate at 3.8% as anticoagulant (BD,
- Vacutainer; Becton, Dickinson and Company, NJ). Blood samples are then
- 87 transported to the Bank of Tissue (Banco de hueso Dr. José E. Gonzalez) where
- by centrifugation at 1800 rpm for 10 minutes (HeraeusMegafuge 1.0R;
- ThermoElectronCorporation) the separation of the 3 layers (White, yellow and red).
- The superior layer rich in plasma will be collected in 50 microliters polypropylene
- 91 tubes (Corning, NY). A final volumen of 16 ml of platelet rich plasma is obtained
- 92 and will transferred to airtight tubes (BD Vacutainer; Becton, Dickinson and
- Company, NJ). The manipulation of the blood samples is made on laminar flow
- cabin biosecurity class II (Logic 3440801; Labconco, KC). The platelet rich plasma
- 95 will be activated with calcium gluconate at 10% (Pisa Farmacéutica, Jalisco,
- 96 México) before using it is placed in the surgical site topically. The PRP simple will
- be divided in two applications, initiating the intervention after the final cuts of the
- 98 TKR components (like the tranexamic acid group).

99 First application: 8 mL of PRP are applied over the surgical site and are left for five 100 minutes then drained out completely by suction. 101 Second application: The rest of the 8 mL are applied over the surgical site after 102 placing the final TKR cemented components (femoral, tibial and patellar), over the 103 surgical site and leaving it without draining. 104 Then a primary closure of the wound is performed (capsule, fascia, subcutaneous 105 tissue and skin) in both groups. A close drainage (Drenovac, NEdren S de R.L. de 106 C.V.) is left intraarticular and fixed to the skin. The drainage will be clamped for 2 107 hours and removed at the 48 hours of the surgery. Thromboprophylaxis (low 108 weight heparin) will be initiated after 6 hours of the end of the surgery. In the 109 postoperative follow up, any patient with hemoglobin levels less than 9mg/dl with 110 anemic syndrome will be transfused. 111 112 References: 113 Levine BR, Haughom B, Strong B, Hellman M, Frank RM. Blood management 114 strategies for total knee arthroplasty. J Am Acad Orthop Surg. 2014 Jun;22(6):361-115 71. doi: 10.5435/JAAOS-22-06-361. Review. PubMed ID: 24860132 116 117 Wind TC, Barfield WR, Moskal JT. The effect of tranexamic acid on blood loss and 118 transfusion rate in primary total knee arthroplasty. J Arthroplasty. 2013 119 Aug;28(7):1080-3. doi: 10.1016/j.arth.2012.11.016. Epub 2013 Mar 28. PubMed

121

122

120

ID: 23541868

Frisch NB, Wessell NM, Charters MA, Yu S, Jeffries JJ, Silverton CD. Predictors

123 and complications of blood transfusion in total hip and knee arthroplasty. J 124 Arthroplasty. 2014 Sep;29(9 Suppl):189-92. doi: 10.1016/j.arth.2014.03.048. Epub 125 2014 May 24. PubMed ID: 25007727 126 127 Moskal JT, Harris RN, Capps SG. Transfusion cost savings with tranexamic acid in 128 primary total knee arthroplasty from 2009 to 2012. J Arthroplasty. 2015 129 Mar;30(3):365-8. doi: 10.1016/j.arth.2014.10.008. Epub 2014 Oct 12. PubMed ID: 130 25458093 131 132 CRASH-2 trial collaborators, Shakur H, Roberts I, Bautista R, Caballero J, Coats T, 133 Dewan Y, El-Sayed H, Gogichaishvili T, Gupta S, Herrera J, Hunt B, Iribhogbe P, 134 Izurieta M, Khamis H, Komolafe E, Marrero MA, Mejía-Mantilla J, Miranda J, 135 Morales C, Olaomi O, Olldashi F, Perel P, Peto R, Ramana PV, Ravi RR, 136 Yutthakasemsunt S. Effects of tranexamic acid on death, vascular occlusive 137 events, and blood transfusion in trauma patients with significant haemorrhage 138 (CRASH-2): a randomised, placebo-controlled trial. Lancet. 2010 Jul 139 3;376(9734):23-32. doi: 10.1016/S0140-6736(10)60835-5. Epub 2010 Jun 14. 140 PubMed ID: 20554319 141 142 Sheth U, Simunovic N, Klein G, Fu F, Einhorn TA, Schemitsch E, Ayeni OR, 143 Bhandari M. Efficacy of autologous platelet-rich plasma use for orthopaedic 144 indications: a meta-analysis. J Bone Joint Surg Am. 2012 Feb 15;94(4):298-307. 145 doi: 10.2106/JBJS.K.00154. Review. PubMed ID: 22241606

146

147 Patel JN, Spanyer JM, Smith LS, Huang J, Yakkanti MR, Malkani AL. Comparison 148 of intravenous versus topical tranexamic acid in total knee arthroplasty: a 149 prospective randomized study. J Arthroplasty. 2014 Aug;29(8):1528-31. doi: 150 10.1016/j.arth.2014.03.011. Epub 2014 Mar 21. PubMed ID: 24768543 151 152 Chimento GF, Huff T, Ochsner JL Jr, Meyer M, Brandner L, Babin S. An evaluation 153 of the use of topical tranexamic acid in total knee arthroplasty. J Arthroplasty. 2013 154 Sep;28(8 Suppl):74-7. doi: 10.1016/j.arth.2013.06.037. PubMed ID: 24034510 155 156 Georgiadis AG, Muh SJ, Silverton CD, Weir RM, Laker MW. A prospective double-157 blind placebo controlled trial of topical tranexamic acid in total knee arthroplasty. J 158 Arthroplasty. 2013 Sep;28(8 Suppl):78-82. doi: 10.1016/j.arth.2013.03.038. Epub 159 2013 Jul 29. PubMed ID: 23906869 160 161 Sarzaeem MM, Razi M, Kazemian G, Moghaddam ME, Rasi AM, Karimi M. 162 Comparing efficacy of three methods of tranexamic acid administration in reducing 163 hemoglobin drop following total knee arthroplasty. J Arthroplasty. 2014 164 Aug;29(8):1521-4. doi: 10.1016/j.arth.2014.02.031. Epub 2014 Mar 6. PubMed ID: 165 24726174 166 167 Alshryda S, Mason J, Sarda P, Nargol A, Cooke N, Ahmad H, Tang S, Logishetty 168 R, Vaghela M, McPartlin L, Hungin AP. Topical (intra-articular) tranexamic acid 169 reduces blood loss and transfusion rates following total hip replacement: a 170 randomized controlled trial (TRANX-H). J Bone Joint Surg Am. 2013 Nov

| 171 | 6;95(21):1969-74. doi: 10.2106/JBJS.L.00908. PubMed ID: 24196467 |
|---|---|
| 172 | |
| 173 | Pace TB, Foret JL, Palmer MJ, Tanner SL, Snider RG. Intraoperative platelet rich |
| 174 | plasma usage in total knee arthroplasty: does it help? ISRN Orthop. 2013 Jul |
| 175 | 28;2013:740173. doi: 10.1155/2013/740173. eCollection 2013. PubMed ID: |
| 176 | 24971180 |
| 177 | |
| 178 | Morishita M, Ishida K, Matsumoto T, Kuroda R, Kurosaka M, Tsumura N. |
| 179 | Intraoperative platelet-rich plasma does not improve outcomes of total knee |
| 180 | arthroplasty. J Arthroplasty. 2014 Dec;29(12):2337-41. doi: |
| 181 | 10.1016/j.arth.2014.04.007. Epub 2014 Apr 13. PubMed ID: 24851794 |
| 182 | |
| 183 | Aggarwal AK, Shashikanth VS, Marwaha N. Platelet-rich plasma prevents blood |
| 184 | loss and pain and enhances early functional outcome after total knee arthroplasty: |
| 185 | a prospective randomised controlled study. Int Orthop. 2014 Feb;38(2):387-95. doi: |
| 186 | 10.1007/s00264-013-2136-6. Epub 2013 Oct 11. PubMed ID: 24114251 |
| 187 | |
| 188 | Bloomfield MR, Klika AK, Molloy RM, Froimson MI, Krebs VE, Barsoum WK. |
| 189 | Prospective randomized evaluation of a collagen/thrombin and autologous platelet |
| 190 | hemostatic agent during total knee arthroplasty. J Arthroplasty. 2012 |
| 191 | May;27(5):695-702. doi: 10.1016/j.arth.2011.09.014. Epub 2011 Oct 27. PubMed |
| 192 | ID: 22035976 |
| 193 | |
| 101 | Gardner M.I. Demetrakonoulos D. Klenchick P.P. Mogar P.A. The efficacy of |

- autologous platelet gel in pain control and blood loss in total knee arthroplasty. An
- analysis of the haemoglobin, narcotic requirement and range of motion. Int Orthop.
- 197 2007 Jun;31(3):309-13. Epub 2006 Jul 1. PubMed ID: 16816947